CLINICAL TRIAL: NCT06339489
Title: Explore the Bone Metabolism Characteristics of Premature Ovarian Insufficiency
Brief Title: The Bone Metabolism Characteristics of Premature Ovarian Insufficiency
Acronym: POI
Status: Recruiting | Type: Observational
Sponsor: Shi Yun (Other)
Responsible Party: Sponsor-Investigator, Shi Yun, Sponsor-Investigator, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Other Study IDs: 2022DZMEC-PG-34
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Premature Ovarian Insufficiency; Bone Diseases, Metabolic; Bone Mineral Density
MeSH Terms: conditions — Primary Ovarian Insufficiency; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POI Group: The patients with premature ovarian insufficiency
  Interventions: Diagnostic Test: Testing the serum levels of bone metabolic markers

INTERVENTIONS:
Diagnostic Test: Testing the serum levels of bone metabolic markers — Testing serum levels of TRACP-5b and BALP, BMD values of lumbar spine L1-L4, left and right hip, left and right femoral neck et.al.

SUMMARY:
Explore the bone metabolism characteristics of premature ovarian insufficiency.

DETAILED DESCRIPTION:
Explore the bone metabolism characteristics of premature ovarian insufficiency, indexes includes serum levels of TRACP-5b and BALP, BMD values of lumbar spine L1-L4, left and right hip, left and right femoral neck et.al.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed by Western medicine with premature ovarian insufficiency. 18 ≤ patients' age ≤ 39 years;. Patients who voluntarily participate in this study, sign an informed consent form.

Exclusion Criteria:

Patients with congenital gonadal dysplasia or a family history similar to "early menopause".

POI patients with acquired organic lesions or ovarian surgery. Patients who have taken Western or herbal medicine artificial cycle therapy or other endocrine therapy in the past three months.

Patients with serious primary diseases and mental disorders such as cardiovascular and cerebrovascular, liver, kidney and hematopoietic system.

Patients who are breastfeeding or pregnant.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biological sex
Study Population: females with premature ovarian insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
tartrate resistant acid phosphatase-5b, TRACP-5b | On the 2~4th day of menstruation (amenorrhea patients are collected when enrolled)
  Blood samples are collected when enrolled.

SECONDARY OUTCOMES:
bone specific alkaline phosphatase, BALP | On the 2~4th day of menstruation (amenorrhea patients are collected when enrolled)
  Blood samples are collected when enrolled.
bone mineral density, BMD | On the 2~4th day of menstruation (amenorrhea patients are collected when enrolled)
  BMD values of lumbar spine L1-L4, left and right hip, left and right femoral neck

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided